CLINICAL TRIAL: NCT00268203
Title: Expanded Access Study of Iodine I 131 Tositumomab for Relapsed/Refractory Low-Grade and Transformed Low-Grade Non-Hodgkin's Lymphoma
Brief Title: Expanded Access Study Of BEXXAR® For Low Grade And Transformed Low-Grade Non-Hodgkin's Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: BEX104545
Record Dates: First submitted 2005-12-20; First posted 2005-12-22 (Estimated); Results first posted 2013-12-09 (Estimated); Last update posted 2017-01-09 (Estimated); Status verified 2016-11

CONDITIONS: Lymphoma, Non-Hodgkin
Keywords: expanded access study; refractory low-grade non-Hodgkin's Lymphoma; Bexxar®; Iodine I 131 Tositumomab; EAP; relapsed low-grade non-Hodgkin's lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin

INTERVENTIONS:
Biological: Iodine I 131 Tositumomab Therapeutic Regimen — Patients will receive unlabeled Tositumomab (450 mg) followed by Tositumomab (35 mg) which has been trace-labeled with 5 mCi of Iodine-131 (dosimetric dose). Whole body counts using a gamma camera will be obtained 3 times between Days 0 and 7 following the dosimetric dose to determine a patient-specific mCi dose of Iodine-131 calculated to deliver the desired total body dose of radiation (either 65 cGy or 75 cGy). The therapeutic dose is administered 7-14 days after the dosimetric dose. Patients will receive unlabeled Tositumomab (450 mg) followed by Tositumomab (35 mg) labeled with the patient-specific dose of Iodine-131 (median dose in previous studies was approximately 85 mCi). Patients who are obese will be dosed based upon 137% of their calculated lean body mass. Patients will be treated with thyroid blocking medication at least 24 hours prior to the dosimetric dose and continuing for 14 days following the therapeutic dose.

SUMMARY:
This is a single arm, multi-center, expanded access study of Iodine I 131 Tositumomab (BEXXAR) therapeutic regimen for patients with relapsed or refractory low-grade or transformed low-grade non-Hodgkin's B-cell lymphoma. The primary objective is to make Iodine I 131 Tositumomab more broadly available to patients. Secondary endpoints will be to obtain additional safety and efficacy information for this treatment regimen. Post study drug administration follow-ups will continue for up to ten years. These will include blood-work and adverse event assessments for 13 weeks post dosing, patient response evaluations at Week 13, Months 6, 12, 18, 24, and Long-Term Follow-ups every 6 months until the elapse of 5 years from the dosimetric dose and then annually thereafter through year 10. Thyroid function will be monitored annually during Long-term follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of low- grade NHL or transformed low-grade NHL (tumor must be CD 20 positive).
* Prior treatment with at least one chemotherapy regimen and have relapsed or progressed, or failed to achieve an objective response on last chemotherapy regimen.
* Karnofsky performance status of at least 60% and anticipated survival of at least 3 months.
* Absolute granulocyte of >/= 1,500/mm3.
* Platelet count of >/= 100,000/mm3, and not require sustained support of hematopoietic cytokines, or transfusion of blood products.
* Adequate renal function (i.e., <1.5x Upper Limit of Normal), and hepatic transaminases (AST <5 times ULN).
* Signed IRB/IEC-approved informed consent.

Exclusion Criteria:

* Patients with a mean of >25% of the intratrabecular marrow space involved with lymphoma.
* Patients who received cytotoxic chemotherapy, radiation therapy, immunotherapy, or cytokine treatment within 4 weeks prior to study entry (6 weeks for nitrosurea compounds) or who exhibit persistent clinical evidence of toxicity.
* Patients who have undergone stem cell or bone marrow transplant, active obstructive hydronephrosis, active infection, New York Heart Association Class III or IV heart disease or other serious illness that would preclude evaluation.
* Known HIV infection.
* Pregnant or nursing patients.
* Patients with prior malignancy other than lymphoma, except for adequately-treated skin cancer, in-situ cervical cancer, or cancer for which the patient has been disease-free for 5 years.
* Patients with progressive disease within 1 year of irradiation arising in a field that has been previously irradiated with more than 3500 cGy.
* Patients who received prior radioimmunotherapy, known brain or leptomeningeal metastases, HAMA positivity.
* Patients who are receiving either approved or non-approved (through another protocol) anti-cancer drugs or biologics.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 765 (Actual)
Dates: Start 1998-09; Primary Completion 2000-03 (Actual); Study Completion 2013-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Annotated Case Report Form: BEX104545 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: BEX104545 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: BEX104545 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: BEX104545 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: NHL=Non-Hodgkin's Lymphoma.
Groups:
- Tositumomab and Iodine I-131 Tositumomab: Participants were treated with a saturated solution of potassium iodide (KI), Lugol's solution, or KI tablets starting at least 24 hours prior to the first infusion of Iodine I-131 Tositumomab (TST) and continuing for 14 days following the last infusion of Iodine I-131 TST. Participants received treatment in two phases. The dosimetric dose was administered in Phase 1 as 450 milligrams (mg) of TST infused over 1 hour (preceded by the administration of oral acetaminophen and an antihistamine), followed by 5 millicurie (mCi) of Iodine I-131 TST infused over 20 minutes (min), followed by a 10-min normal saline flush. The therapeutic dose, administered 7-14 days after the dosimetric dose, was administered as 450 mg of TST infused over 1 hour (preceded by the administration of oral acetaminophen and an antihistamine), followed by the appropriate activity (mCi) of Iodine I-131 TST infused over 20 min, followed by a 10-min normal saline flush.
Period: Overall Study
Arm/Group | Tositumomab and Iodine I-131 Tositumomab
Started | 765
Completed 2 Years of Follow-up | 62
Completed | 118 (These participants completed 10 years of follow-up.)
Not Completed | 647
Not completed — Lost to Follow-up | 92
Not completed — Withdrawal by Subject | 9
Not completed — Received Other NHL Therapy | 7
Not completed — Progressive Disease | 359
Not completed — Death | 84
Not completed — Reason Not Specified | 34
Not completed — Completed 2 Years of Follow-up | 62

BASELINE CHARACTERISTICS:
Arm/Group | Tositumomab and Iodine I-131 Tositumomab
Number analyzed (Participants) | 765
Age, Continuous [Mean (Standard Deviation); unit: Years] | 58.8 (11.5)
Gender [Count of Participants; unit: Participants]
  Female | 354
  Male | 411
Race/Ethnicity, Customized [Number; unit: participants] — Race data were not collected; ethnicity data were collected and are presented instead.
  participants
    White | 711
    Hispanic | 19
    Asian | 7
    Black | 20
    Native American | 1
    Portuguese | 1
    Middle Eastern | 1
    Iranian | 1
    Indian | 2
    Arab | 1
    Peruvian | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Unconfirmed Response (Complete Response or Partial Response) and Unconfirmed Complete Response
Description: A participant was defined as a responder if he/she sustained a complete response (CR: the disappearance of all detectable clinical and radiographic evidence of disease and all disease-related symptoms) or partial response (PR: greater than or equal to a 50% decrease in the sum of the product of perpendicular diameter [SPPD] determined at Baseline; no increase in the size of the other nodes, liver, or spleen; no new sites of disease). Response was evaluated by an investigator per guidelines developed by The International Workshop to Standardize Response Criteria for Non-Hodgkin's Lymphoma.
Time Frame: From randomization until the first documented complete response or partial response (up to 161 months)
Population: Intent-to-Treat (ITT) Population: participants receiving any study drug. Only those participants evaluable for unconfirmed response (those with at least one response assessment) were analyzed.
Measure: Number; unit: Participants
Arm/Group | Tositumomab and Iodine I-131 Tositumomab
Number analyzed (Participants) | 746
Participants
  CR or PR | 437
  CR | 238

2. Primary Outcome: Number of Participants With Confirmed Response (Complete Response or Partial Response) and Confirmed Complete Response
Description: A participant was defined as a responder if he/she sustained a complete response (CR: the disappearance of all detectable clinical and radiographic evidence of disease and all disease-related symptoms) or partial response (PR: greater than or equal to a 50% decrease in the sum of the product of perpendicular diameter [SPPD] determined at Baseline; no increase in the size of the other nodes, liver, or spleen; no new sites of disease). Response was evaluated by an investigator per guidelines developed by The International Workshop to Standardize Response Criteria for Non-Hodgkin's Lymphoma. A confirmed response (CR and PR) requires that the response be confirmed by another response (same or better) at least 4 weeks apart.
Time Frame: From randomization until the first documented complete response or partial response (up to 161 months)
Population: Intent-to-Treat (ITT) Population: participants receiving any study drug. Only those participants evaluable for confirmed response (those with at least one response assessment) were analyzed.
Measure: Number; unit: Participants
Arm/Group | Tositumomab and Iodine I-131 Tositumomab
Number analyzed (Participants) | 502
Participants
  CR or PR | 339
  CR | 196

3. Primary Outcome: Duration of Response for Participants With Unconfirmed Response (CR+PR)
Description: Duration of response is defined as the time from the first documented CR (the disappearance of all detectable clinical and radiographic evidence of disease and all disease-related symptoms) or PR (greater than or equal to a 50% decrease in the SPPD determined at Baseline; no increase in the size of the other nodes, liver, or spleen; no new sites of disease) until disease progression (PD). PD is defined as greater than or equal to a 50% increase from nadir in the SPPD for all measurable disease. Lesion changes believed to represent measurement variation associated with radiographic technique should not be classified as PD. Response was evaluated by an investigator per guidelines developed by the International Workshop to Standardize Response Criteria for Non-Hodgkin's Lymphoma.
Time Frame: From the time of the first documented response (CR or PR) until disease progression (up to 161 months)
Population: ITT Population. Only those participants with an unconfirmed CR or PR were analyzed for duration of unconfirmed response. Participants who did not have disease progression were censored in the analysis at the date of their last contact.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Tositumomab and Iodine I-131 Tositumomab
Number analyzed (Participants) | 437
Months | 21.0 [17.3 to NA] — The upper limit of the confidence interval could not be calculated because there were too few events of progression.

4. Primary Outcome: Duration of Response for Participants With Confirmed Response (CR+PR)
Description: Duration of response is defined as the time from the first documented CR (the disappearance of all detectable clinical and radiographic evidence of disease and all disease-related symptoms) or PR (greater than or equal to a 50% decrease in the SPPD determined at Baseline; no increase in the size of the other nodes, liver, or spleen; no new sites of disease) until disease progression (PD). PD is defined as greater than or equal to a 50% increase from nadir in the SPPD for all measurable disease. Lesion changes believed to represent measurement variation associated with radiographic technique should not be classified as PD. Response was evaluated by an investigator per guidelines developed by the International Workshop to Standardize Response Criteria for Non-Hodgkin's Lymphoma. A confirmed response (CR and PR) requires that the response be confirmed by another response (same or better) at least 4 weeks apart.
Time Frame: From the time of the first documented response (CR or PR) until disease progression (up to 161 months)
Population: ITT Population. Only those participants with a confirmed CR or PR were analyzed for duration of confirmed response. Participants who did not have disease progression were censored in the analysis at the date of their last contact.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Tositumomab and Iodine I-131 Tositumomab
Number analyzed (Participants) | 339
Months | NA [NA to NA] — A median cannot be calculated because the survival distribution from the Kaplan-Meier survival curve does not reach 50%.

5. Primary Outcome: Duration of Response (DOR) in Unconfirmed Complete Responders
Description: DOR is defined as the time from the first documented response to the first documented disease progression. Unconfirmed CR is defined as the disappearance of all detectable clinical and radiographic evidence of disease and all disease-related symptoms. Response was evaluated by an investigator per guidelines developed by The International Workshop to Standardize Response Criteria for Non-Hodgkin's Lymphoma.
Time Frame: From the time of the first documented unconfirmed CR until PD (up to 161 months)
Population: ITT Population. Only those participants with an unconfirmed CR were included in this analysis of duration of response. Participants who did not have disease progression were censored in the analysis at the date of their last contact.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Tositumomab and Iodine I-131 Tositumomab
Number analyzed (Participants) | 238
Months | NA [NA to NA] — A median cannot be calculated because the survival distribution from the Kaplan-Meier survival curve does not reach 50%.

6. Primary Outcome: Duration of Response (DOR) in Confirmed Complete Responders
Description: DOR is defined as the time from the first documented response to the first documented disease progression. CR is defined as the disappearance of all detectable clinical and radiographic evidence of disease and all disease-related symptoms. A confirmed response (CR and PR) requires that the response be confirmed by another response (same or better) at least 4 weeks apart.
Time Frame: From the time of the first documented CR until PD (up to 161 months)
Population: ITT Population. Only those participants with a confirmed CR were included in this analysis of duration of response. Participants who did not have disease progression were censored in the analysis at the date of their last contact.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Tositumomab and Iodine I-131 Tositumomab
Number analyzed (Participants) | 196
Months | NA [NA to NA] — A median cannot be calculated because the survival distribution from the Kaplan-Meier survival curve does not reach 50%.

7. Primary Outcome: Time to Progression or Death
Description: Time to progression is defined as the time from the treatment start date to the first documented incidence of disease progression (PD) or death. PD is defined as greater than or equal to a 50% increase from nadir in the SPPD for all measurable disease. Lesion changes believed to represent measurement variation associated with radiographic technique should not be classified as PD.
Time Frame: From the treatment start date to the first documented incidence of disease progression (PD) or death (up to 161 months)
Population: ITT Population. Participants who did not have disease progression or death were censored in the analysis at the date of their last contact.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Tositumomab and Iodine I-131 Tositumomab
Number analyzed (Participants) | 765
Months | 9.2 [6.8 to 10.8]

8. Secondary Outcome: Time to Treatment Failure
Description: Time to treatment failure is defined as the time from the date of the dosimetric dose to the first occurrence of the following: treatment withdrawal, decision to seek additional therapy, study removal, disease progression, receipt of alternative therapy for lymphoma, or death study withdrawal for any reason. Participants withdrawn for reasons other than progression or death were censored at their date of withdrawal.
Time Frame: From the dosimetric dose to the first occurrence of the following: treatment withdrawal, decision to seek additional therapy, study removal, disease progression, receipt of alternative therapy, or death (up to 161 months)
Population: ITT Population. Participants who did not experience treatment failure were censored at the date of their last contact.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Tositumomab and Iodine I-131 Tositumomab
Number analyzed (Participants) | 765
Months | 9.0 [6.3 to 10.4]

ADVERSE EVENTS:
Arm/Group | Tositumomab and Iodine I-131 Tositumomab
Serious Adverse Events (participants affected / at risk) | 204/765
Other Adverse Events (participants affected / at risk) | 650/765
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tositumomab and Iodine I-131 Tositumomab (N=765)
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 34
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 18
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Central nervous system lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Endometrial cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Hodgkin's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Infected neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastases to breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Neuroendocrine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Neuroendocrine carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Non-Hodgkin's lymphoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Rectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Refractory cytopenia with unilineage dysplasi (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Richter's syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Salivary gland cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Tongue neoplasm malignant stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Anaemia (Blood and lymphatic system disorders) | 16
Thrombocytopenia (Blood and lymphatic system disorders) | 16
Pancytopenia (Blood and lymphatic system disorders) | 10
Febrile neutropenia (Blood and lymphatic system disorders) | 9
Neutropenia (Blood and lymphatic system disorders) | 9
Leukopenia (Blood and lymphatic system disorders) | 5
Bone marrow failure (Blood and lymphatic system disorders) | 1
Granulocytopenia (Blood and lymphatic system disorders) | 1
Haemolytic anaemia (Blood and lymphatic system disorders) | 1
Lymphadenitis (Blood and lymphatic system disorders) | 1
Pneumonia (Infections and infestations) | 8
Sepsis (Infections and infestations) | 8
Cellulitis (Infections and infestations) | 4
Abdominal abscess (Infections and infestations) | 1
Bronchitis (Infections and infestations) | 1
Cellulitis orbital (Infections and infestations) | 1
Clostridium difficile colitis (Infections and infestations) | 1
Device related sepsis (Infections and infestations) | 1
Herpes zoster (Infections and infestations) | 1
Infection (Infections and infestations) | 1
Kidney infection (Infections and infestations) | 1
Neutropenic sepsis (Infections and infestations) | 1
Peritoneal abscess (Infections and infestations) | 1
Pneumonia respiratory syncytial viral (Infections and infestations) | 1
Pseudomonal sepsis (Infections and infestations) | 1
Skin bacterial infection (Infections and infestations) | 1
Staphylococcal sepsis (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Urosepsis (Infections and infestations) | 1
Pyrexia (General disorders) | 19
Chills (General disorders) | 6
Asthenia (General disorders) | 3
Fatigue (General disorders) | 3
Pain (General disorders) | 3
Chest pain (General disorders) | 2
Oedema peripheral (General disorders) | 2
Generalised oedema (General disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 10
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 6
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 4
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Hydropneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
Laryngeal obstruction (Respiratory, thoracic and mediastinal disorders) | 1
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 1
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 1
Stridor (Respiratory, thoracic and mediastinal disorders) | 1
Nausea (Gastrointestinal disorders) | 6
Vomiting (Gastrointestinal disorders) | 6
Abdominal pain (Gastrointestinal disorders) | 3
Diarrhoea (Gastrointestinal disorders) | 3
Constipation (Gastrointestinal disorders) | 2
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2
Abdominal pain upper (Gastrointestinal disorders) | 1
Abdominal wall mass (Gastrointestinal disorders) | 1
Ascites (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 1
Haematemesis (Gastrointestinal disorders) | 1
Intestinal obstruction (Gastrointestinal disorders) | 1
Intestinal perforation (Gastrointestinal disorders) | 1
Odynophagia (Gastrointestinal disorders) | 1
Oesophagitis (Gastrointestinal disorders) | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1
Umbilical hernia (Gastrointestinal disorders) | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 9
Hypercalcaemia (Metabolism and nutrition disorders) | 5
Cachexia (Metabolism and nutrition disorders) | 1
Decreased appetite (Metabolism and nutrition disorders) | 1
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1
Lactic acidosis (Metabolism and nutrition disorders) | 1
Tumour lysis syndrome (Metabolism and nutrition disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 6
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5
Myalgia (Musculoskeletal and connective tissue disorders) | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1
Atrial fibrillation (Cardiac disorders) | 2
Cardiac failure congestive (Cardiac disorders) | 2
Supraventricular tachycardia (Cardiac disorders) | 2
Tachycardia (Cardiac disorders) | 2
Atrioventricular block complete (Cardiac disorders) | 1
Cardio-respiratory arrest (Cardiac disorders) | 1
Left ventricular failure (Cardiac disorders) | 1
Pericardial effusion (Cardiac disorders) | 1
Sinus bradycardia (Cardiac disorders) | 1
Ventricular tachycardia (Cardiac disorders) | 1
Spinal cord compression (Nervous system disorders) | 2
Cerebrovascular accident (Nervous system disorders) | 1
Convulsion (Nervous system disorders) | 1
Depressed level of consciousness (Nervous system disorders) | 1
Lethargy (Nervous system disorders) | 1
Paralysis (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Transient ischaemic attack (Nervous system disorders) | 1
VIIth nerve paralysis (Nervous system disorders) | 1
Renal failure acute (Renal and urinary disorders) | 3
Renal failure (Renal and urinary disorders) | 2
Ureteric obstruction (Renal and urinary disorders) | 2
Dysuria (Renal and urinary disorders) | 1
Confusional state (Psychiatric disorders) | 3
Mental disorder due to a general medical condition (Psychiatric disorders) | 1
Mental status changes (Psychiatric disorders) | 1
Neutrophil count decreased (Investigations) | 2
Clostridium test positive (Investigations) | 1
Haemoglobin decreased (Investigations) | 1
Weight decreased (Investigations) | 1
Hypotension (Vascular disorders) | 2
Deep vein thrombosis (Vascular disorders) | 1
Haemorrhage (Vascular disorders) | 1
Bile duct obstruction (Hepatobiliary disorders) | 1
Hepatic lesion (Hepatobiliary disorders) | 1
Hyperthyroidism (Endocrine disorders) | 1
Serum sickness (Immune system disorders) | 1
Pelvic fracture (Injury, poisoning and procedural complications) | 1
Ulna fracture (Injury, poisoning and procedural complications) | 1
Acute febrile neutrophilic dermatosis (Skin and subcutaneous tissue disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tositumomab and Iodine I-131 Tositumomab (N=765)
Absolute neutrophil count < 1000 cells/mm^3 (Investigations) | 293
Platelets < 50000 cells/mm^3 (Investigations) | 278
White blood cells < 2000 cells/mm^3 (Investigations) | 260
Hemoglobin < 8.0 grams per deciliter (Investigations) | 91
Fatigue (General disorders) | 166
Pyrexia (General disorders) | 82
Chills (General disorders) | 57
Oedema peripheral (General disorders) | 23
Pain (General disorders) | 19
Asthenia (General disorders) | 13
Influenza like illness (General disorders) | 13
Chest pain (General disorders) | 12
Chest discomfort (General disorders) | 11
Malaise (General disorders) | 6
Feeling hot (General disorders) | 5
Axillary pain (General disorders) | 2
Discomfort (General disorders) | 2
Face oedema (General disorders) | 2
Feeling cold (General disorders) | 2
Local swelling (General disorders) | 2
Oedema (General disorders) | 2
Crepitations (General disorders) | 1
Feeling abnormal (General disorders) | 1
Infusion site pain (General disorders) | 1
Infusion site pruritus (General disorders) | 1
Injection site haematoma (General disorders) | 1
Local reaction (General disorders) | 1
Mucosal inflammation (General disorders) | 1
Sensation of foreign body (General disorders) | 1
Spinal pain (General disorders) | 1
Thirst (General disorders) | 1
Nausea (Gastrointestinal disorders) | 135
Vomiting (Gastrointestinal disorders) | 52
Diarrhoea (Gastrointestinal disorders) | 49
Abdominal pain (Gastrointestinal disorders) | 26
Constipation (Gastrointestinal disorders) | 17
Abdominal discomfort (Gastrointestinal disorders) | 12
Stomatitis (Gastrointestinal disorders) | 12
Abdominal distension (Gastrointestinal disorders) | 9
Dyspepsia (Gastrointestinal disorders) | 7
Dysphagia (Gastrointestinal disorders) | 6
Abdominal pain upper (Gastrointestinal disorders) | 5
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 4
Gingival bleeding (Gastrointestinal disorders) | 4
Dry mouth (Gastrointestinal disorders) | 3
Epigastric discomfort (Gastrointestinal disorders) | 3
Melaena (Gastrointestinal disorders) | 3
Oral pain (Gastrointestinal disorders) | 3
Rectal haemorrhage (Gastrointestinal disorders) | 3
Abdominal pain lower (Gastrointestinal disorders) | 2
Flatulence (Gastrointestinal disorders) | 2
Haematochezia (Gastrointestinal disorders) | 2
Mouth ulceration (Gastrointestinal disorders) | 2
Oedema mouth (Gastrointestinal disorders) | 2
Toothache (Gastrointestinal disorders) | 2
Abdominal tenderness (Gastrointestinal disorders) | 2
Ascites (Gastrointestinal disorders) | 1
Cheilitis (Gastrointestinal disorders) | 1
Faces discoloured (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Gastrointestinal pain (Gastrointestinal disorders) | 1
Gingival pain (Gastrointestinal disorders) | 1
Glossodynia (Gastrointestinal disorders) | 1
Haematemesis (Gastrointestinal disorders) | 1
Haemorrhoids (Gastrointestinal disorders) | 1
Hiatus hernia (Gastrointestinal disorders) | 1
Intestinal obstruction (Gastrointestinal disorders) | 1
Intra-abdominal haemorrhage (Gastrointestinal disorders) | 1
Lip dry (Gastrointestinal disorders) | 1
Lip pain (Gastrointestinal disorders) | 1
Lip swelling (Gastrointestinal disorders) | 1
Oesophagitis (Gastrointestinal disorders) | 1
Oral disorder (Gastrointestinal disorders) | 1
Oral pruritus (Gastrointestinal disorders) | 1
Paraesthesia oral (Gastrointestinal disorders) | 1
Regurgitation (Gastrointestinal disorders) | 1
Tongue disorder (Gastrointestinal disorders) | 1
Anaemia (Blood and lymphatic system disorders) | 97
Thrombocytopenia (Blood and lymphatic system disorders) | 60
Neutropenia (Blood and lymphatic system disorders) | 51
Pancytopenia (Blood and lymphatic system disorders) | 9
Leukopenia (Blood and lymphatic system disorders) | 7
Febrile neutropenia (Blood and lymphatic system disorders) | 6
Granulocytopenia (Blood and lymphatic system disorders) | 4
Lymph node pain (Blood and lymphatic system disorders) | 4
Lymphadenopathy (Blood and lymphatic system disorders) | 4
Bone marrow failure (Blood and lymphatic system disorders) | 2
Microcytic anaemia (Blood and lymphatic system disorders) | 1
Priritus (Skin and subcutaneous tissue disorders) | 45
Rash (Skin and subcutaneous tissue disorders) | 37
Urticaria (Skin and subcutaneous tissue disorders) | 22
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 20
Night sweats (Skin and subcutaneous tissue disorders) | 17
Erythema (Skin and subcutaneous tissue disorders) | 9
Rash generalised (Skin and subcutaneous tissue disorders) | 4
Rash macular (Skin and subcutaneous tissue disorders) | 4
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 3
Dermatitis (Skin and subcutaneous tissue disorders) | 3
Petechiae (Skin and subcutaneous tissue disorders) | 3
Skin efoliation (Skin and subcutaneous tissue disorders) | 3
Ecchymosis (Skin and subcutaneous tissue disorders) | 2
Pruritus generalised (Skin and subcutaneous tissue disorders) | 2
Rash erythematous (Skin and subcutaneous tissue disorders) | 2
Skin disorder (Skin and subcutaneous tissue disorders) | 2
Skin lesion (Skin and subcutaneous tissue disorders) | 2
Swelling face (Skin and subcutaneous tissue disorders) | 2
Acne (Skin and subcutaneous tissue disorders) | 1
Blood blister (Skin and subcutaneous tissue disorders) | 1
Dermal cyst (Skin and subcutaneous tissue disorders) | 1
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1
Exfoliative rash (Skin and subcutaneous tissue disorders) | 1
Leukocytoclastic vasculitis (Skin and subcutaneous tissue disorders) | 1
Leukoplakia (Skin and subcutaneous tissue disorders) | 1
Livedo reticularis (Skin and subcutaneous tissue disorders) | 1
Penile ulceration (Skin and subcutaneous tissue disorders) | 1
Rash pruritic (Skin and subcutaneous tissue disorders) | 1
Skin irritation (Skin and subcutaneous tissue disorders) | 1
Umbilical erythema (Skin and subcutaneous tissue disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 55
Myalgia (Musculoskeletal and connective tissue disorders) | 39
Back pain (Musculoskeletal and connective tissue disorders) | 25
Pain in extremity (Musculoskeletal and connective tissue disorders) | 15
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 9
Bone pain (Musculoskeletal and connective tissue disorders) | 7
Muscle spasms (Musculoskeletal and connective tissue disorders) | 7
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 6
Groin pain (Musculoskeletal and connective tissue disorders) | 5
Muscular weakness (Musculoskeletal and connective tissue disorders) | 4
Neck pain (Musculoskeletal and connective tissue disorders) | 4
Flank pain (Musculoskeletal and connective tissue disorders) | 3
Joint stiffness (Musculoskeletal and connective tissue disorders) | 2
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 2
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 2
Pain in jaw (Musculoskeletal and connective tissue disorders) | 2
Sensation of heaviness (Musculoskeletal and connective tissue disorders) | 2
Arthritis (Musculoskeletal and connective tissue disorders) | 1
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 1
Mobility decreased (Musculoskeletal and connective tissue disorders) | 1
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 41
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 39
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 17
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 14
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 8
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 8
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 7
Productive cough (Respiratory, thoracic and mediastinal disorders) | 7
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 6
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 6
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 4
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 4
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 3
Pharyngeal oedema (Respiratory, thoracic and mediastinal disorders) | 3
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 3
Throat tightness (Respiratory, thoracic and mediastinal disorders) | 3
Dry throat (Respiratory, thoracic and mediastinal disorders) | 2
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 2
Oropharyngeal discomfort (Respiratory, thoracic and mediastinal disorders) | 2
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 2
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 2
Wheezing (Respiratory, thoracic and mediastinal disorders) | 2
Allergic cough (Respiratory, thoracic and mediastinal disorders) | 1
Apnoea (Respiratory, thoracic and mediastinal disorders) | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1
Nasal ulcer (Respiratory, thoracic and mediastinal disorders) | 1
Orthopnoea (Respiratory, thoracic and mediastinal disorders) | 1
Painful respiration (Respiratory, thoracic and mediastinal disorders) | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1
Rales (Respiratory, thoracic and mediastinal disorders) | 1
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1
Stridor (Respiratory, thoracic and mediastinal disorders) | 1
Headache (Nervous system disorders) | 53
Dizziness (Nervous system disorders) | 34
Somnolence (Nervous system disorders) | 15
Dysgeusia (Nervous system disorders) | 11
Hypoaesthesia (Nervous system disorders) | 11
Paraesthesia (Nervous system disorders) | 6
Burning sensation (Nervous system disorders) | 3
Peripheral sensory neuropathy (Nervous system disorders) | 3
Lethargy (Nervous system disorders) | 2
Migraine (Nervous system disorders) | 2
Syncope (Nervous system disorders) | 2
Akathisia (Nervous system disorders) | 1
Aphonia (Nervous system disorders) | 1
Balance disorder (Nervous system disorders) | 1
Dysarthria (Nervous system disorders) | 1
Loss of consciousness (Nervous system disorders) | 1
Memory impairment (Nervous system disorders) | 1
Peripheral motor neuropathy (Nervous system disorders) | 1
Peroneal nerve palsy (Nervous system disorders) | 1
Restless legs syndrome (Nervous system disorders) | 1
Sciatica (Nervous system disorders) | 1
Sensory loss (Nervous system disorders) | 1
Sinus headache (Nervous system disorders) | 1
Tremor (Nervous system disorders) | 1
VIIth nerve paralysis (Nervous system disorders) | 1
Upper respiratory tract infection (Infections and infestations) | 20
Sinusitis (Infections and infestations) | 14
Pneumonia (Infections and infestations) | 13
Herpes zoster (Infections and infestations) | 10
Urinary tract infection (Infections and infestations) | 8
Oral herpes (Infections and infestations) | 6
Influenza (Infections and infestations) | 5
Nasopharyngitis (Infections and infestations) | 5
Rhinitis (Infections and infestations) | 4
Bronchitis (Infections and infestations) | 3
Cellulitis (Infections and infestations) | 3
Herpes virus infection (Infections and infestations) | 2
Oral candidiasis (Infections and infestations) | 2
Otitis media (Infections and infestations) | 2
Tooth abscess (Infections and infestations) | 2
Tooth infection (Infections and infestations) | 2
Vaginal infection (Infections and infestations) | 2
Wound infection (Infections and infestations) | 2
Abscess oral (Infections and infestations) | 1
Bronchitis viral (Infections and infestations) | 1
Candidiasis (Infections and infestations) | 1
Chronic sinusitis (Infections and infestations) | 1
Conjunctivitis infective (Infections and infestations) | 1
Ear infection (Infections and infestations) | 1
Genital herpes (Infections and infestations) | 1
Herpes simplex (Infections and infestations) | 1
Hordeolum (Infections and infestations) | 1
Infection (Infections and infestations) | 1
Lower respiratory tract infection (Infections and infestations) | 1
Paronychia (Infections and infestations) | 1
Parotitis (Infections and infestations) | 1
Pharyngitis (Infections and infestations) | 1
Varicella (Infections and infestations) | 1
Vulvovaginal mycotic infection (Infections and infestations) | 1
Haemoglobin decreased (Investigations) | 19
Weight decreased (Investigations) | 13
Platelet count decreased (Investigations) | 8
White blood cell count decreased (Investigations) | 6
Blood pressure systolic decreased (Investigations) | 4
Body temperature increased (Investigations) | 4
Neutrophil count decreased (Investigations) | 3
Blood creatinine increased (Investigations) | 2
Blood thyroid stimulating hormone increased (Investigations) | 2
Haematocrit decreased (Investigations) | 2
Red blood cell count decreased (Investigations) | 2
Band neutrophil count decreased (Investigations) | 1
Blood pressure increased (Investigations) | 1
Blood test abnormal (Investigations) | 1
Electroencephalogram abnormal (Investigations) | 1
Heart rate irregular (Investigations) | 1
Prostatic specific antigen increased (Investigations) | 1
Urine output decreased (Investigations) | 1
Urine output increased (Investigations) | 1
Hypothyroidism (Endocrine disorders) | 44
Goitre (Endocrine disorders) | 2
Hyperthyroidism (Endocrine disorders) | 2
Thyroid disorder (Endocrine disorders) | 2
Thyroid pain (Endocrine disorders) | 1
Thyroiditis (Endocrine disorders) | 1
Decreased appetite (Metabolism and nutrition disorders) | 36
Dehydration (Metabolism and nutrition disorders) | 6
Hyperglycaemia (Metabolism and nutrition disorders) | 4
Hyperkalaemia (Metabolism and nutrition disorders) | 3
Hypercalcaemia (Metabolism and nutrition disorders) | 2
Hypophagia (Metabolism and nutrition disorders) | 2
Cachexia (Metabolism and nutrition disorders) | 1
Failure to thrive (Metabolism and nutrition disorders) | 1
Hyperlipidaemia (Metabolism and nutrition disorders) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1
Malnutrition (Metabolism and nutrition disorders) | 1
Hypotension (Vascular disorders) | 16
Flushing (Vascular disorders) | 11
Hypertension (Vascular disorders) | 5
Hot flush (Vascular disorders) | 3
Deep vein thrombosis (Vascular disorders) | 2
Pallor (Vascular disorders) | 2
Peripheral coldness (Vascular disorders) | 2
Haemorrhage (Vascular disorders) | 1
Orthostatic hypotension (Vascular disorders) | 1
Phlebitis (Vascular disorders) | 1
Insomnia (Psychiatric disorders) | 10
Confusional state (Psychiatric disorders) | 7
Depression (Psychiatric disorders) | 6
Anxiety (Psychiatric disorders) | 4
Disorientation (Psychiatric disorders) | 1
Panic attack (Psychiatric disorders) | 1
Diplopia (Eye disorders) | 4
Vision blurred (Eye disorders) | 4
Eye pain (Eye disorders) | 3
Ocular hyperaemia (Eye disorders) | 3
Photophobia (Eye disorders) | 3
Conjunctivitis (Eye disorders) | 2
Eye pruritus (Eye disorders) | 2
Eye swelling (Eye disorders) | 2
Eyelid oedema (Eye disorders) | 2
Lacrimation increased (Eye disorders) | 2
Visual impairment (Eye disorders) | 2
Abnormal sensation in eye (Eye disorders) | 1
Dark circles under eyes (Eye disorders) | 1
Eye irritation (Eye disorders) | 1
Eyelid ptosis (Eye disorders) | 1
Vitreous floaters (Eye disorders) | 1
Contusion (Injury, poisoning and procedural complications) | 9
Foot fracture (Injury, poisoning and procedural complications) | 2
Arthropod bite (Injury, poisoning and procedural complications) | 1
Excoriation (Injury, poisoning and procedural complications) | 1
Fall (Injury, poisoning and procedural complications) | 1
Ligament injury (Injury, poisoning and procedural complications) | 1
Ligament sprain (Injury, poisoning and procedural complications) | 1
Procedural pain (Injury, poisoning and procedural complications) | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 1
Tracheal deviation (Injury, poisoning and procedural complications) | 1
Wrist fracture (Injury, poisoning and procedural complications) | 1
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4
Tumour flare (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
Lymphoma transformation (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Follicle centre lymphoma, follicular grade I, II, III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Intraductal proliferative breast lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Pollakiuria (Renal and urinary disorders) | 4
Renal failure (Renal and urinary disorders) | 3
Dysuria (Renal and urinary disorders) | 2
Bladder discomfort (Renal and urinary disorders) | 1
Bladder spasm (Renal and urinary disorders) | 1
Haematuria (Renal and urinary disorders) | 1
Hydronephrosis (Renal and urinary disorders) | 1
Micturition urgency (Renal and urinary disorders) | 1
Nocturia (Renal and urinary disorders) | 1
Ureteric obstruction (Renal and urinary disorders) | 1
Urinary incontinence (Renal and urinary disorders) | 1
Urinary retention (Renal and urinary disorders) | 1
Pelvic pain (Reproductive system and breast disorders) | 3
Vaginal haemorrhage (Reproductive system and breast disorders) | 2
Breast induration (Reproductive system and breast disorders) | 1
Erectile dysfunction (Reproductive system and breast disorders) | 1
Genital rash (Reproductive system and breast disorders) | 1
Menorrhagia (Reproductive system and breast disorders) | 1
Scrotal oedema (Reproductive system and breast disorders) | 1
Testicular pain (Reproductive system and breast disorders) | 1
Testicular swelling (Reproductive system and breast disorders) | 1
Vaginal discharge (Reproductive system and breast disorders) | 1
Vulvovaginal pruritus (Reproductive system and breast disorders) | 1
Tachycardia (Cardiac disorders) | 4
Palpitation (Cardiac disorders) | 2
Ventricular extrasystoles (Cardiac disorders) | 2
Arrthythmia (Cardiac disorders) | 1
Bradycardia (Cardiac disorders) | 1
Cardiac failure congestive (Cardiac disorders) | 1
Left ventricular dysfunction (Cardiac disorders) | 1
Sinus bradycardia (Cardiac disorders) | 1
Sinus tachycardia (Cardiac disorders) | 1
Ventricular tachycardia (Cardiac disorders) | 1
Ear discomfort (Ear and labyrinth disorders) | 2
Tinnitus (Ear and labyrinth disorders) | 2
Ear congestion (Ear and labyrinth disorders) | 1
Ear pain (Ear and labyrinth disorders) | 1
Hearing impaired (Ear and labyrinth disorders) | 1
Otorrhoea (Ear and labyrinth disorders) | 1
Vertigo (Ear and labyrinth disorders) | 1
Hypersensitivity (Immune system disorders) | 4
Anaphylactoid reaction (Immune system disorders) | 2
Hypogammaglobulinaemia (Immune system disorders) | 1
Thyroid therapy (Surgical and medical procedures) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.